CLINICAL TRIAL: NCT03704805
Title: Effect of a Psychological Intervention on Antiretroviral Therapy Outcomes and Symptoms of Common Mental Disorders in HIV-positive Adults in Rural Zimbabwe
Brief Title: Effect of a Psychological Intervention on Antiretroviral Therapy and Mental Health Outcomes in HIV-positive Adults in Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: SolidarMed (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FB-ART
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Mental Disorder; HIV Infections
MeSH Terms: conditions — Mental Disorders; HIV Infections

STUDY DESIGN:
Intervention Model Description: Cluster-randomized, controlled, two-arm multicenter, superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-Solving Therapy (Experimental): Participants in the intervention group receive the friendship bench intervention in addition to all services provided according to enhanced standard of care.
  Interventions: Behavioral: Friendship bench intervention; Other: Enhanced Standard of Care
- Enhanced Standard of Care (Active Comparator): Participants in the control group receive enhanced standard of care.
  Interventions: Other: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: Friendship bench intervention — The friendship bench intervention consists of six individual counseling sessions and a peer-led group activity. Individual counseling is based on problem-solving therapy and delivered by lay health workers. During individual counseling, participants will be actively encouraged to identify and tackle problems leading to sub-optimal antiretroviral therapy adherence. In the group activity, participants are taught an income generating skill and have the opportunity to share personal experience with former participants of the intervention.
  Arms: Problem-Solving Therapy
Other: Enhanced Standard of Care — Study participants receive information on available routine services for common mental disorders, a nurse-led brief support counseling, assessment for antidepressant medication (fluoxetine) by the clinic nurse, and referral to a psychiatric facility if needed, in addition to the standard of care provided according to national antiretroviral therapy guidelines.

SUMMARY:
The aim of the study is to examine the effect of a psychological intervention on antiretroviral therapy outcomes and symptoms of common mental health disorders among adults living with HIV and common mental disorders in rural Zimbabwe.

DETAILED DESCRIPTION:
Common mental disorders are highly prevalent among people living with HIV. Left untreated, common mental disorders cause substantial disability and undermine individuals' ability to adhere to antiretroviral therapy, leading to poor antiretroviral therapy outcomes.

A recent cluster-randomized controlled trial from Harare, Zimbabwe showed that the friendship bench intervention (i.e. six sessions of problem-solving therapy delivered by lay health workers followed by a peer support group) effectively reduced symptoms of common mental disorders, but the effect of the intervention on antiretroviral therapy outcomes and its effectiveness in the rural setting has not been studied.

To examine the effect of the friendship bench intervention on antiretroviral therapy outcomes and symptoms of common mental disorders among adults living with HIV and common mental disorders in rural Zimbabwe, a cluster-randomized trial is conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Use of first-line antiretroviral therapy for at least 6 months
* Resident in Bikita District
* Knowledge of English or Shona language
* Ability to comprehend the information on the study
* Positive screening for common mental disorders (SSQ-14 score ≥9)
* Providing informed consent

Exclusion Criteria:

* Current psychosis / cognitive impairment
* Clinical AIDS (WHO clinical stage 4)
* Known pregnancy or ≤3 months postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Average difference in mean antiretroviral therapy adherence between 2 and 6 months | 2-6 months
  Adherence will be calculated as percentage of prescribed doses taken and measured with the Medication Event Monitoring System (MEMS)

SECONDARY OUTCOMES:
Difference in mean antiretroviral therapy adherence between 1 and 12 months | 1-12 months
  Adherence will be calculated as percentage of prescribed doses taken and measured with the Medication Event Monitoring System (MEMS)
Difference in change from baseline in Shona Symptoms Questionnaire (SSQ-14) score | At month 3, 6, 9, and 12
  The Shone Symptoms Questionnaire is a 14 item tool. The reported total score is between 0 and 14. 14 is the highest level of mental disorder. Each item adds a score of 0 or 1 to the total score.
Difference in change from baseline in Patient Health Questionnaire (PHQ-9) score | At month 3, 6, 9, and 12
  The Patient Health Questionnaire is a 9 item tool. The reported total score is between 0 and 27. 27 is the highest level of depression. Each item adds a score of 0 to 3 to the total score.
Viral load suppression (<1000 copies per milliliter) | At month 6 (i.e., day 180 ± 90 days) and month 12 (i.e., day 360 ± 90 days)
  Categorical (yes, no, invalid or missing).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas D Haas, PhD, Principal Investigator — Institute of Social and Preventive Medicine (ISPM), University of Bern; Cordelia Kunzekwenyika, MD, Principal Investigator — SolidarMed, Swiss Organisation for Health in Africa
Locations (1):
- Solidarmed, Masvingo, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haas AD, Kunzekwenyika C, Manzero J, Hossmann S, Limacher A, van Dijk JH, Manhibi R, von Groote P, Hobbins MA, Verhey R, Egger M; Friendship Bench ART trial group. Effect of the Friendship Bench Intervention on Antiretroviral Therapy Outcomes and Mental Health Symptoms in Rural Zimbabwe: A Cluster Randomized Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2323205. doi: 10.1001/jamanetworkopen.2023.23205. PMID 37440230
- [Derived] Haas AD, Kunzekwenyika C, Manzero J, Hossmann S, Limacher A, van Dijk JH, Manhibi R, von Groote P, Hobbins MA, Verhey R, Egger M; Friendship Bench ART trial group. Effect of the Friendship Bench intervention on antiretroviral therapy outcomes and mental health symptoms in rural Zimbabwe: A cluster randomized trial. medRxiv [Preprint]. 2023 Jan 22:2023.01.21.23284784. doi: 10.1101/2023.01.21.23284784. PMID 36711671
- [Derived] Haas AD, Kunzekwenyika C, Hossmann S, Manzero J, van Dijk J, Manhibi R, Verhey R, Limacher A, von Groote PM, Manda E, Hobbins MA, Chibanda D, Egger M; IeDEA Southern Africa. Symptoms of common mental disorders and adherence to antiretroviral therapy among adults living with HIV in rural Zimbabwe: a cross-sectional study. BMJ Open. 2021 Jul 7;11(7):e049824. doi: 10.1136/bmjopen-2021-049824. PMID 34233999